CLINICAL TRIAL: NCT07403916
Title: Influence of Age on the Choice of Treatment and Prognosis in Patients With Resectable Gastric Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: P. Herzen Moscow Oncology Research Institute (Other Government)
Responsible Party: Principal Investigator, Vakhtang Begiashvili, PhD student, P. Herzen Moscow Oncology Research Institute
Other Study IDs: 129
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Gastric Cancer (GC); Next-generation Sequencing; Molecular Analysis
Keywords: Gastric cancer surgery; Next-generation sequencing; Gastric cancer treatment
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Уoung-adult age group: age 18-44 yr.
  Interventions: Diagnostic Test: Next-generation sequencing
- Middle-aged group: age 45-59 yr.
  Interventions: Diagnostic Test: Next-generation sequencing
- Eldery age group: age 60-74 yr.
  Interventions: Diagnostic Test: Next-generation sequencing
- Senior age group: age > 75 yr.
  Interventions: Diagnostic Test: Next-generation sequencing

INTERVENTIONS:
Diagnostic Test: Next-generation sequencing — Technology for determining the sequence of DNA to study genetic variation associated with diseases or other biological phenomena

SUMMARY:
Next-generation sequencing (NGS) and biomarkers play a key role in the diagnosis and personalized therapy of gastric cancer. These technologies provide a deep understanding of the molecular basis of the disease.

NGS allows simultaneous analysis of multiple genes, identifying mutations and changes in their expression. In case of stomach cancer, this makes it possible to identify specific mutations to determine prognosis and treatment choice, study the genomic profiles of patients to find targets for targeted and immunotherapy.

The use of NGS and biomarkers allows the development of individualized treatment regimens, increasing effectiveness and reducing side effects. Biomarker analysis also helps to track the progression of the disease and identify patients at high risk of relapse.

The study of molecular genetic markers in tumor tissues, as well as the influence of genetic and age-related factors, is an important scientific and clinical task. Solving this problem will create a personalized approach to patient management.

This work examines the influence of age on the choice of treatment tactics and prognosis in patients with resectable gastric cancer. The main focus is on the analysis of surgical, chemotherapeutic, topographic, pathomorphological, and molecular genetic correlations in various age groups.

DETAILED DESCRIPTION:
Gastric cancer remains one of the most important malignant tumors with significant geographical and regional differences in prevalence. Despite the decrease in the incidence of gastric cancer in advanced economies, this pathology still ranks fifth among patients with malignant neoplasms. As for cancer mortality rates, stomach cancer ranks third. Stomach cancer continues to be one of the most significant oncological diseases in the world, ranking fifth in terms of prevalence according to global statistics from GLOBOCAN 2022.

Modern medicine uses diagnostic technology - Next-generation sequencing (NGS), and biomarkers play an important role in the diagnosis, prognosis, and treatment of stomach cancer. These technologies provide a deep understanding of the molecular mechanisms underlying the disease and open up new possibilities for personalized therapy. NGS allows simultaneous analysis of multiple genes and detection of mutations, changes in gene expression and other genetic features. In the context of stomach cancer, next-generation sequencing allows for identification of mutations: Detection of specific mutations associated with stomach cancer can help determine prognosis and select appropriate treatment, study of the genomic profiles of patients: To identify potential targets for therapy, including immune and targeted drugs.

With the help of NGS and biomarkers, doctors can develop individualized treatment regimens for different age groups, which increases the effectiveness of therapy and reduces side effects. Biomarker analysis allows you to track the progression of cancer and identify patients with a high risk of recurrence. The study and determination of molecular genetic markers in tumor tissues, as well as the analysis of genetic and age-related factors influencing the development of gastric cancer, is an important scientific and clinical task. Solving this problem may allow us to develop a personalized approach to patient management.

This scientific paper will address the issue of the influence of age on the choice of treatment tactics and prognosis in patients with resectable gastric cancer. The main focus is on surgical, chemotherapeutic, topographic, pathomorphological, and molecular genetic correlations of various age groups in resectable gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed diagnosis of gastric cancer
* The resectable stage of the disease (I-III)
* Availability of complete clinical data, including age, gender, stage of the disease, concomitant diseases, treatment tactics and outcomes
* Indicated radical surgical intervention both at the first stage and after neoadjuvant chemotherapy
* Localization of the tumor: Type II-III cardioesophageal junction according to Siewert, upper, middle and lower third of the body, angle of the stomach or antrum (U,M,L-level according to the Japanese classification)

Exclusion Criteria:

* The presence of metastases in distant organs at the time of diagnosis
* Primary-multiple tumors
* Diagnostic and palliative surgery
* Incomplete clinical data
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with clinically documented primary gastric cancer undergoing elective surgery with curative intent
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 months

SECONDARY OUTCOMES:
Mutational burden and genomic instability features assessed by NGS | 3 months
Spectrum of somatic mutations identified by NGS | 3 months
Disease free survival | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrey Ryabov, MD, PhD, Study Director — P.Herzen Moscow Oncological Research Institute; Vakhtang Begiashvili, PhD student, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Vladimir Khomyakov, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Nadezhda Volchenko, MD, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute; Shatalov Peter, PhD, Principal Investigator — P.Herzen Moscow Oncological Research Institute
Locations (1):
- P.Herzen Moscow Oncological Research Institute, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided